CLINICAL TRIAL: NCT03752515
Title: A Chinese Registry to Determine the Genetics Risk Factors and Serumal Biomarkers for Acute Coronary Syndrome
Brief Title: A Registry Study on Genetics and Biomarkers of Acute Coronary Syndrome
Acronym: ARSGB-ACS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Beijing Institute of Heart, Lung and Blood Vessel Diseases (Other)
Responsible Party: Sponsor
Other Study IDs: BeijingIHLBVD2018010
Record Dates: First submitted 2018-10-31; First posted 2018-11-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Coronary Artery Disease; Acute Coronary Syndrome; Acute Myocardial Infarction; Unstable Angina
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome; Angina, Unstable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — If a blood specimen is obtained, it will be separated and stored at -80 ℃ as plasma, viable cells, and extracted DNA. If a saliva specimen is obtained, it is stored for DNA.
  If a tissue specimen is obtained, it will be cut into small pieces and stored at liquid nitrogen.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- case-ACS-MACE: ACS patients with poor prognosis
- control-ACS-MACE: ACS patients with good prognosis
- Health-control: general population without ACS

SUMMARY:
This is a national registry study to determine genetics risk factors and serial biomarkers of Acute Coronary Syndrome.

ELIGIBILITY:
ACS Case Inclusion Criteria:

* Written informed consent has been provided.
* Contact Order Form has been provided.
* Aged 18 years or older.
* Hospitalized within 48 hours of onset of symptoms.
* Diagnosis of STEMI, NSTEMI or UA using the following definitions:

  1.Criteria for STEMI diagnosis:
  1. History of chest pain/discomfort and
  2. Persistent ST-segment elevation (> 30 min) of ≥ 0.1 mV in 2 or more contiguous ECG leads or presumed new left bundle branch block (LBBB) on admission and
  3. Elevation of cardiac biomarkers (CK-MB, troponins): at least one value above the 99th percentile of the local laboratory upper reference limit.

  2.Criteria for NSTEMI diagnosis:

  1.History of chest pain/discomfort and 2.Lack of persistent ST-segment elevation, LBBB or intraventricular conduction disturbances and 3.Elevation of cardiac biomarkers (CK-MB, troponins): at least one value above the 99th percentile of the local laboratory upper reference limit. 3.Criteria for Unstable Angina diagnosis:
  1. Symptoms of angina at rest or on minimal exercise and
  2. At least 0.5mm ST deviation in at least 2 leads and
  3. No increase in biomarkers of necrosis
  4. OR objective evidence of ischaemia by non-invasive imaging OR significant coronary stenosis as determined by the treating physician at angiography if this is standard practice in study site.

     Case Exclusion Criteria:

     Patients will not be eligible to participate if any of the following exclusion criteria are present:
* UA, STEMI and NSTEMI precipitated by or as a complication of surgery, trauma, or GI bleeding or post-PCI.
* UA, STEMI and NSTEMI occurring in patients already hospitalized for other reasons.
* Presence of any condition/circumstance which in the opinion of the investigator could significantly limit the complete follow up of the patient (e.g. tourist, non-native speaker or does not understand the local language, psychiatric disturbances).
* Presence of serious/severe co-morbidities in the opinion of the investigator which may limit short term (i.e. 6 month) life expectancy.
* Current participation in a randomised interventional clinical trial.

Control Inclusion Criteria:

* Age and gender are matched with cases.
* No Coronary Artery Disease was detected by Coronary CT examination.
* Normal biochemical indicators.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Case-ACS-MACE group consists of patients who was diagnosed as Acute Coronary Syndrome and had a poor prognosis during follow up.
  Control-ACS-MACE group consists of patients who was diagnosed as Acute Coronary Syndrome and had a good prognosis during follow up.
  Health control group is general population without Acute Coronary Syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2015-06-02 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Age for each participant | These data is collected from the cases' medical record in an average of 1 month after the sample recruiting
  current age and onset age
Gender for each participant | These data is collected from the cases' medical record in an average of 1 month after the sample recruiting
  male or female
Height for each participant | These data is collected from the cases' medical record in an average of 1 month after the sample recruiting
  cm cm cm
Weight for each participant | These data is collected from the cases' medical record in an average of 1 month after the sample recruiting
  kg
Contact information for each participant | These data is collected from the cases' medical record in an average of 1 month after the sample recruiting
  telephone
Past Medical History | These data is collected from the cases' medical record in an average of 1 month after the sample recruiting
  including disease history, surgical history, and medical history
Lifestyle | These data is collected from the cases' medical record in an average of 1 month after the sample recruiting
  including smoking history and drinking, specify how many years smoking or drinking lasted and detail quantity per day
Biochemical | These data is collected from the cases' medical record in an average of 1 month after the sample recruiting
  including blood lipid, fasting glucose, Creatinine and so on
Biomarkers | These data is collected from the cases' medical record in an average of 1 month after the sample recruiting
  including cTnI, BNP, hs-CRP, and so on
Overall lesion profiles | These data is collected from the cases' medical record in an average of 1 month after the sample recruiting
  how many vessels involved
Echocardiography | These data is collected from the cases' medical record in an average of 1 month after the sample recruiting
  LVEF and so on
Medication at discharge | These data is collected from the cases' medical record in an average of 1 month after the sample recruiting
Genetic data | Sequencing will be carried out in an average of 3 months after sample recruiting
  Exon sequencing data or genotypes of candidate SNPs
Metabolomic profile on Liquid Chromatograph Mass Spectrometer/Mass Spectrometer analysis of serum sample. | The data is collected from lab in an average of 3 month after the sample recruiting
  The results of metabolomics will be measured by mass spectrometry, including lipids, sugars, amino acids, carnitine, choline, arachidonic acid, sterol and free fat acid . All of metabolites will be quantitative (unit: mol/L). Identification of molecules via Human Metabolites Database will be reported online.
Detection of miRNAs expression in each participant using the qRT-PCT method. | The data is collected from lab in an average of 3 month after the sample recruiting
  Relative expression levels of miRNA were analyzed using the 2-△Ct method and U6 was used as an endogenous control.
Detection of candidate biomarkers in each participant using proteome detection or ELASA | The data is collected from lab in an average of 12 month after the sample recruiting
Major adverse cardiovascular events (MACE) in overall population, defined as composite of all-cause death, Heart Failure, recurrent myocardial infarction, stroke or ischemia-driven revascularization. | These data is collected during follow-up visit after discharge
  HF includes in-hospital and long-term post-discharge HF incidence

CONTACTS AND LOCATIONS:
Overall Officials: Jie Du, PHD, Study Director — Beijing Anzhen Hospital
Locations (6):
- China (6):
  - Beijing Anzhen Hospital, Beijing
  - Beijing Luhe Hospital, Capital Medical University, Beijing
  - The First Affiliated Hospital of Dalian Medical University, Dalian
  - The Second Hospital of Dalian Medical University, Dalian
  - The First Hospital of Jilin University, Jilin
  - People's Hospital of Henan University, Zhengzhou

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ma J, Ma K, Chen J, Yang X, Gao F, Gao H, Zhang H, Ma XL, Du J, Li P, Li Y. Development and Validation of Risk Stratification for Heart Failure After Acute Coronary Syndrome Based on Dynamic S100A8/A9 Levels. J Am Heart Assoc. 2025 Feb 4;14(3):e037401. doi: 10.1161/JAHA.124.037401. Epub 2025 Feb 3. PMID 39895550
- [Derived] Li Y, Chen B, Yang X, Zhang C, Jiao Y, Li P, Liu Y, Li Z, Qiao B, Bond Lau W, Ma XL, Du J. S100a8/a9 Signaling Causes Mitochondrial Dysfunction and Cardiomyocyte Death in Response to Ischemic/Reperfusion Injury. Circulation. 2019 Aug 27;140(9):751-764. doi: 10.1161/CIRCULATIONAHA.118.039262. Epub 2019 Jun 21. PMID 31220942